CLINICAL TRIAL: NCT07289932
Title: "Clinical Evaluation of Self-Assembling Peptides Versus Tri-Calcium Phosphate Based Varnish in Treatment of White Spot Lesions; Split-Mouth Randomized Clinical Trial"
Acronym: SAP VS TCP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OPD 22 24 (D)
Record Dates: First submitted 2025-12-05; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: White Spot Lesions
Keywords: White spot lesions Orthodontic white spot lesions Enamel demineralization Enamel remineralization; P11-4 Curodont Repair Tri-calcium phosphate varnish; Biomimetic remineralization Split-mouth randomized controlled tria
MeSH Terms: interventions — tenocyclidine

STUDY DESIGN:
Intervention Model Description: "This is a split-mouth randomized controlled clinical trial. Each participant will receive the self-assembling peptide varnish (Curodont Repair) on one side of the mouth and the tri-calcium phosphate varnish (Clinpro White Varnish) on the contralateral side, allowing within-patient comparison."
Who Masked: Participant, Outcomes Assessor
Masking Description: "This study uses a double-blind split-mouth design. Participants and outcome assessors are blinded to the intervention allocation. The treating clinician cannot be blinded due to product differences in application, but will not be involved in outcome evaluation. Data analysis will be performed with blinded group coding."
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curodont Repair (Self-Assembling Peptide, SAP P11-4) (Experimental): Application of Curodont Repair varnish to eligible white spot lesions on one side of the mouth at baseline and after 3 months.
  Interventions: Other: Curodont Repair (SAP P11-4)
- Clinpro White Varnish (Tri-Calcium Phosphate, TCP) (Active Comparator): Application of Clinpro White Varnish to eligible white spot lesions on the contralateral side of the mouth at baseline and after 3 months.
  Interventions: Other: Clinpro White Varnish (Tri-Calcium Phosphate, TCP)

INTERVENTIONS:
Other: Curodont Repair (SAP P11-4) — Application of Curodont Repair, a self-assembling peptide (P11-4) varnish designed to penetrate subsurface enamel lesions and promote hydroxyapatite formation. The varnish will be applied to eligible white spot lesions on one side of the anterior teeth at baseline and re-applied after 3 months according to manufacturer's instructions."
  Arms: Curodont Repair (Self-Assembling Peptide, SAP P11-4)
Other: Clinpro White Varnish (Tri-Calcium Phosphate, TCP) — "Application of Clinpro White Varnish containing tri-calcium phosphate and fluoride, designed to deliver bioavailable calcium, phosphate, and fluoride ions to the enamel surface. The varnish will be applied to eligible white spot lesions on the contralateral side of the anterior teeth at baseline and re-applied after 3 months according to manufacturer's instructions."
  Arms: Clinpro White Varnish (Tri-Calcium Phosphate, TCP)

SUMMARY:
Brief Summary:

This randomized controlled clinical trial will evaluate the effectiveness of two remineralizing agents in the treatment of white spot lesions (WSLs) in young adults. White spot lesions are early signs of enamel demineralization that commonly develop after orthodontic treatment. The study will compare a self-assembling peptide-based varnish (Curodont Repair, SAP P11-4) with a tri-calcium phosphate-based varnish (Clinpro White Varnish, 3M) using a split-mouth design.

A total of patients aged 15-25 years with at least one eligible WSL on each side of the anterior teeth will be enrolled. Each patient will receive Curodont Repair on one side and Clinpro White Varnish on the contralateral side. Treatments will be applied at baseline and repeated after 3 months. Lesions will be evaluated using standardized digital photography, ICDAS II scoring, lesion size measurements, and patient satisfaction questionnaires at baseline, 3, 6, and 9 months.

The primary outcome is the change in color of white spot lesions over 9 months. Secondary outcomes include changes in lesion size, ICDAS scores, and patient-reported satisfaction. The study is double-blinded (patients and outcome assessors) and conducted at the Faculty of Dentistry, Ain Shams University.

DETAILED DESCRIPTION:
White spot lesions (WSLs) represent the earliest clinically detectable stage of enamel caries and are a common consequence of fixed orthodontic treatment. These lesions are characterized by increased opacity of enamel due to subsurface demineralization. Conventional fluoride-based strategies can promote surface remineralization but often fail to achieve full penetration into the lesion body, limiting complete enamel repair.

Novel biomimetic approaches, such as self-assembling peptides (SAP P11-4), have been developed to address this limitation. SAP molecules can diffuse into the subsurface lesion and form a three-dimensional scaffold that attracts calcium and phosphate ions from saliva, facilitating de novo hydroxyapatite formation and deeper remineralization. In contrast, tri-calcium phosphate (TCP) varnishes provide bioavailable minerals in combination with fluoride to enhance surface remineralization.

Although both strategies show promising laboratory and clinical results, there is limited evidence directly comparing their clinical performance in patients with orthodontically induced WSLs. This study aims to fill that gap by using a split-mouth, randomized controlled design to compare the effectiveness of Curodont Repair (SAP P11-4) and Clinpro White Varnish (TCP) in young adult patients.

The study will focus on the extent of remineralization as assessed by digital imaging and color analysis, supplemented by changes in lesion size and ICDAS II scoring. Patient satisfaction will also be evaluated to capture subjective outcomes of esthetic improvement. Findings from this study are expected to contribute to evidence-based recommendations for minimally invasive management of WSLs.

ELIGIBILITY:
Inclusion Criteria:

- A minimum of one tooth affected by early carious lesions (ICDAS-II codes 1 or 2) in both sides of the mouth that do not require invasive treatment.

* Age 15 years and ≤ 25 years
* Size and form of the carious lesions must both be fully visible, and accessible
* Willing and able to attend the on-study visits and to observe good oral hygiene throughout the study
* Provide written informed consent before participation in the study as subjects were minors, informed consent will provided by the parent and/or legal guardian.
* patients not on medication affecting their salivary flow and medically free (ASA class I).

Exclusion Criteria:

* Evidence of tooth erosion.

  * any form of fluoride application before the study treatment.
  * patients with hypoplastic enamel defects, multiple restorations on the facial surfaces.
  * High caries risk patients

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in color of white spot lesions | Baseline, 3 months, 6 months, and 9 months
  "Change in color and appearance of white spot lesions will be assessed using standardized digital intraoral photography and eLAB color analysis system. The color difference (ΔE) values will be calculated to quantify remineralization."

SECONDARY OUTCOMES:
Change in lesion size | Baseline, 3 months, 6 months, and 9 months
  "Lesion size will be measured from standardized digital photographs using ImageJ software to calculate changes in lesion surface area."

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR